CLINICAL TRIAL: NCT03921112
Title: Role of Lung Ultrasound in Weaning From Mechanical Ventilation in Postoperative Neurosurgical ICU Patients :Prospective , Randomized Double-blinded Study
Brief Title: Role of Lung Ultrasound in Weaning From Mechanical Ventilation in Postoperative Neurosurgical ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R26/2019
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Intensive Care (ICU)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lung ultrasound (Active Comparator)
  Interventions: Device: lung ultrasound; Other: routine tools
- x-ray, ABG, RSBI, Vetilator parameters (Active Comparator)
  Interventions: Other: routine tools

INTERVENTIONS:
Device: lung ultrasound — bedside lung ultrasound will be done for patients
  Arms: lung ultrasound
Other: routine tools — chest X-ray , ABG, RSBI, Ventilator parameters will be done for all patients

SUMMARY:
The aim of this study is to demonstrate the role of lung ultrasound in weaning from mechanical ventilation in neurosurgical ICU patients compared to the ordinary tools as chest X-ray , ABG, rapid shallow breathing index, ventilator parameters.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients
* ASAI ,ASAII, ASAIII

Exclusion Criteria:

* Patients or gurdians refuse
* Patients with pneumthorax
* Patients with pleural effusion
* Patients with surgical emphysema
* Glasco coma score more than 8
* Patients on high inotropic support
* patients with diaphragmatic paralysis

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
success of weaning | success of weaning for 48 hours
  trans-thoracic lung ultrasound will be done to patients to start weaning

CONTACTS AND LOCATIONS:
Overall Officials: Amin m Alansary, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt